CLINICAL TRIAL: NCT05991726
Title: Taking an Active Role in Your Own Healthcare: A Delphi Survey for Key Stakeholders to Identify Priority Self-management Outcomes for Chronic Kidney Disease (SM-CKD Delphi Study)
Brief Title: A Delphi Survey for Key Stakeholders to Identify Priority Self-management Outcomes for Chronic Kidney Disease
Status: Completed | Type: Observational
Sponsor: University of Leicester (Other)
Responsible Party: Sponsor
Other Study IDs: 33721
Record Dates: First submitted 2023-08-07; First posted 2023-08-15 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Chronic Kidney Diseases
Keywords: Survey; Chronic Kidney disease; Stakeholder
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Professional Expert: This includes Healthcare professionals (HCPs) who look after people with CKD in the UK, anyone involved in designing, developing, managing and commissioning of CKD healthcare in the UK and researchers interested in self-management or CKD
  Interventions: Other: Other: Survey
- Cohort 2: Non-Professional Expert: People living with a diagnosis of CKD. This survey focusses on people with non-dialysis CKD, typically stages 3-4. However, this study does not exclude participation by those at a more advanced stage or receiving renal replacement therapy (dialysis or transplant) as these people also have lived experience of earlier stages to draw on. This will also include 'significant others' whom are supporters or carers of people with CKD such as a family member or a partner of a person with CKD.
  Interventions: Other: Other: Survey

INTERVENTIONS:
Other: Other: Survey — Multiple survey rounds identifying most important outcomes for effective self-management for non-dialysis CKD

SUMMARY:
The purpose of this Delphi study is to identify priority outcomes for self-management in earlier (non-dialysis) stages of CKD from the perspectives of different stakeholder groups in the UK. The findings of this study will be used to inform outcome measure selection for research and clinical evaluations of self-management resources and to support implementation, commissioning and uptake.

DETAILED DESCRIPTION:
Chronic Kidney Disease (CKD) is a progressive condition affecting more than 1.8 million people in England

Effective self-management is important for people living with CKD like many Long-Term Conditions. Self-management in its broadest term can be summarised as individuals participating in the day-to-day management of their chronic condition

Theory- and evidence-based tools and resources for self-management education and support are required to encourage health-promoting behaviours. However, outcomes valued by key stakeholders are necessary to ensure robust evaluation in research settings and clinical practice

A Delphi study is carried out to generate consensus on outcomes that are valued by the stakeholder groups in this study. The Delphi study will undergo 3-4 survey rounds

Adult CKD patient participants living in the UK and their significant others were recruited via social media adverts shared by our research team and English kidney community organisations. Healthcare professionals, commissioners and policymakers (professional groups) based in the UK were recruited by direct email invitations to our extensive contacts in the field

ELIGIBILITY:
Inclusion Criteria:

* People with diagnosis of CKD in the UK
* Their close family and friend
* Healthcare professionals who look after people with CKD in the UK
* Anyone involved in designing, developing, managing and commissioning CKD healthcare services in the UK
* Researchers related in a topic related to self-management or CKD

Exclusion Criteria:

* Any participant residing outside of the UK

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. People living with CKD. This survey focusses on people with non-dialysis CKD, typically stages 3-4. However, we will not exclude participation by those at a more advanced stage or receiving renal replacement therapy (dialysis or transplant) as these people also have lived experience of earlier stages to draw on.
  2. Carers and Supporters of people with CKD (expected to be a significant other i.e. spouse or partner, close family member or friend that are involved in the regular care and support to a person living with CKD)
  3. Healthcare professionals (HCPs) who look after people with CKD in the UK
  4. Anyone involved in designing, developing, managing and commissioning of CKD healthcare in the UK
  5. Researchers interested in self-management or CKD
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2022-05-05 (Actual); Primary Completion 2023-04-03 (Actual); Study Completion 2023-04-03 (Actual)

PRIMARY OUTCOMES:
Open ended free text question | Between 3 to 6 month
  Round 1- Participants are asked to describe the 3 most important outcomes for self-management in people with non-dialysis CKD from their own perspective or opinion
Consensus Rating | Between 3 to 6 month
  Round 2- Participants are asked to rate each item on a 9 point Likert-type scale, the lowest scoring items are removed (consensus is predefined as ≥ 70% on each item scoring on the critical importance scale that is a score of 7-9).
Consensus Ranking | Between 3 to 6 month
  Round 3- Participants are asked to rank each item and themes in order from high to low importance to identify the most valued outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- University of Leicester, Leicester, United Kingdom